CLINICAL TRIAL: NCT02937649
Title: Multicentric Randomized Prospective Study Assessing the Impact of the Bougie Calibration Size During Laparoscopic Sleeve Gastrectomy on the Rate of Postoperative Staple-line Leak Rate
Brief Title: Bougie Sleeve Trial
Acronym: BOUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P150933
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Morbid Obesity
Keywords: Obesity; Bariatric surgery; Sleeve gastrectomy; Staple-line Leak; Bougie; Calibration
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic sleeve gastrectomy using 48-Fr bougie (Experimental): Patients will undergo laparoscopic sleeve gastrectomy with a 48-Fr (16 mm) bougie
  Interventions: Procedure: Laparoscopic sleeve gastrectomy using 48-Fr bougie
- Laparoscopic sleeve gastrectomy using standard care bougie (Active Comparator): Patients will undergo laparoscopic sleeve gastrectomy with a standard care bougie (34, 36 or 38-Fr)
  Interventions: Procedure: Laparoscopic sleeve gastrectomy using standard care bougie

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy using 48-Fr bougie — After gastric mobilization, the 48-Fr bougie is inserted through the mouth by the anesthesiologist and positioned in the stomach. Patient is blind to the type of bougie used. Gastrectomy is performed alongside the calibration bougie.
  Arms: Laparoscopic sleeve gastrectomy using 48-Fr bougie
Procedure: Laparoscopic sleeve gastrectomy using standard care bougie — After gastric mobilization, the standard care bougie is inserted through the mouth by the anesthesiologist and positioned in the stomach. Patient is blind to the type of bougie used. Gastrectomy is performed alongside the calibration bougie.
  Arms: Laparoscopic sleeve gastrectomy using standard care bougie

SUMMARY:
Staple-line leak is the most frequent and incapacitating complication after laparoscopic sleeve gastrectomy (LSG). The aim of this prospective randomized trial is to compare the staple-line leak rate after LSG according to the use of a standard bougie calibre (34, 36 or 38 Fr) or 48-Fr, assuming that a higher diameter is correlated with a lower risk of leak, without lowering long-term weight loss.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (LSG) has become an increasing bariatric procedure. The most common complication is gastric leak from the staple line, observed in approximately 3% of cases, and can result in long and incapacitating treatment. The diameter of the bougie used to calibrate the remnant stomach could impact the rate of gastric leak, a higher diameter being correlated with a lower risk of leak, without lowering long-term weight loss.

The aim of this prospective randomized trial is to compare the outcomes of LSG according to the use of a standard care bougie calibre or 48-Fr on postoperative gastric leak and mid-term weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years
* Sleeve gastrectomy as a primary bariatric procedure
* Body Mass Index (BMI) > 40 kg/m² or > 35 kg/m² associated with at least one comorbidity susceptible to improve after surgery (including arterial hypertension, obstructive sleep apnea syndrome and other severe respiratory disorders, severe metabolic disorders, particularly type 2 diabetes, incapacitating osteo-articular disorders, non alcoholic steatohepatitis)
* Decision for intervention after multidisciplinary discussion
* Written informed consent

Exclusion Criteria:

* Previous upper abdominal surgery (cholecystectomy excepted)
* ASA (American Society of Anesthesiologists) score > 3
* Ongoing pregnancy or breast feeding
* Esophagus pathology or disorder (esophageal varices, esophageal diverticula, esophageal tumors, esophageal strictures)
* Coagulation disorder
* Patient not covered by social security service and patient on AME
* Patient under legal guardianship and trusteeship
* Patient with known silicon allergy (calibration bougie contains medical silicon)
* More generally, all other contraindications to the use of esophageal bougie MID-TUBE that have been the subject of a scientific paper or have been identified by the practitioner or practitioners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1658 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2025-06-08 (Estimated); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative gastric leak rate | 30 days following the procedure
  Postoperative gastric leak rate during the first month following the procedure will be proven either on:
  * Morphologic examination (with contrast ingestion)
  * Blue dye test during surgical reintervention or postoperative course
  * Contrast opacification during endoscopy

SECONDARY OUTCOMES:
Postoperative morbidity rate | 90 days following the procedure
  Postoperative morbidity rate will be calculated regarding any complication occurring 90 days following the procedure.
Short-term weight loss | At 3 and 6 months after the procedure
  Short-term weight loss will be assessed by calculation of excess weight loss at 3 and 6 months after the procedure.
Mid-term weight loss | At 1 and 2 years after the procedure
  Mid-term weight loss will be assessed by calculation of excess weight loss at 1 and 2 years after the procedure.
Quality of life related to health | At 3 months, 6 months, 1 year and 2 years after the procedure
  Quality of life related to health will be assessed at 3 months, 6 months, 1 year and 2 years after the procedure with the validated GIQLI scale (Gastro Intestinal Quality of Life Index)

CONTACTS AND LOCATIONS:
Overall Officials: Hadrien TRANCHART, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Côte de Nacre CHU de Caen, Caen
  - CHU Antoine Béclère, Clamart
  - Centre hospitalier Intercommunal de Créteil, Créteil
  - Hôpital MICHALLON, CHU de Grenoble, La Tronche
  - Hôpital Dupuytren - Limoges, Limoges
  - Clinique de l'Yvette, Longjumeau
  - Service de chirurgie générale et digestive, œsogastrique et bariatrique - Hôpital Bichat, Paris
  - CHI - Centre Hospitalier Poissy/Saint-Germain-en-Laye, Poissy
  - CH Saint-Denis, Saint-Denis
  - Clinique Mutualiste Chirurgicale, Saint-Etienne
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaillard M, Lainas P, Agostini H, Dagher I, Tranchart H. Impact of the calibration bougie diametre during laparoscopic sleeve gastrectomy on the rate of postoperative staple-line leak (BOUST): study protocol for a multicentre randomized prospective trial. Trials. 2021 Nov 15;22(1):806. doi: 10.1186/s13063-021-05734-3. PMID 34781991